CLINICAL TRIAL: NCT00495885
Title: Efficacy and Safety of 2 mg/Day of M100907 on Sleep Maintenance Insomnia With a Sub-study of the Effect of M100907 on Stable Type II Diabetes Mellitus: a 12-week, Multi-center, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of M100907 on Sleep Maintenance Insomnia With a Sub-study in Stable Type II Diabetes Mellitus
Acronym: SAMS12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTE6672; Eudract: 2006-006677-25
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep problems; insomnia; sleeplessness; primary insomnia; insomnia disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — volinanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volinanserin (Experimental): Volinanserin 2 mg for a maximum of 87 days
  Interventions: Drug: volinanserin (M100907)
- Placebo (Placebo Comparator): Placebo for volinanserin for a maximum of 106 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: volinanserin (M100907) — oral, one tablet taken around bedtime
  Arms: Volinanserin
Drug: Placebo — oral, one tablet taken around bedtime
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess efficacy and safety of volinanserin in the population of patients complaining of sleep maintenance insomnia. The objective of the substudy is to assess glycemic control in the subgroup of patients with type II diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) criteria
* Disturbances of sleep maintenance criteria based on patient's information related to sleep pattern during the preceding month

Sub-study :

* Patients will be included if they have an established medical diagnosis of type II Diabetes Mellitus, and have been treated either with an oral hypoglycemic agent and/or insulin for at least three months prior to the Screening Visit (with stable regimen for at least one month prior to screening)

Exclusion Criteria:

* Females who are lactating or who are pregnant
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* Consumption of xanthine-containing beverages (i.e. tea, coffee, cola) comprising more than 5 cups/day
* Participation in another trial having received study medication within 1 month before the screening visit
* Body Mass Index ≥ 33
* Use of over-the-counter medications such as tryptophan, valerian root, kava, melatonin, St. John's Wort, Alluna or prescription sleep medication
* Use of any substance with psychotropic effects or properties know to affect sleep/wake
* History of primary hypersomnia, narcolepsy, breathing-related sleep disorder, circadian rhythm sleep disorder, parasomnia, dyssomnia
* Clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder
* Positive qualitative urine drug screen (opiates, cocaine, amphetamine…)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
change from baseline to 12 weeks for Sleep Maintenance Insomnia using patient reported Wake After Sleep Onset (pr-WASO) | 12 weeks

SECONDARY OUTCOMES:
Change from baseline to 12-week of "General Productivity" domain from Functional Outcomes of Sleep Questionnaire (FOSQ). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)